CLINICAL TRIAL: NCT06494995
Title: The Combination of AK104 and Low-dose Radiation Therapy in Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma After Failure of First-line Systemic Therapy: a Phase II Study
Brief Title: AK104 and Low-dose Radiation in Recurrent/Metastatic HNSCC After Failure of First-line Systemic Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu Wang, Professor, M.D., Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDRT-ICB 1.0; 2312288-4 (Other: Institutional Review Board)
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: low-dose radiotherapy; low-dose radiation; cadonilimab; CTLA-4; PD-1; Stereotactic Body Radiation Therapy; Hybrid radiation; Immune modulation
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Radiotherapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid RT (Experimental): Patients will receive treatment of low-dose radiotherapy and cadonilimab, combined with selective lesions stereotactic radiotherapy.
  Interventions: Drug: Cadonilimab; Radiation: Low-dose radiotherapy; Radiation: SBRT
- Metronomic chemotherapy and LDRT (Experimental): Patients will receive treatment of low-dose radiotherapy and cadonilimab, combined with capecitabine metronomic chemotherapy.
  Interventions: Drug: Cadonilimab; Radiation: Low-dose radiotherapy; Drug: Capecitabine

INTERVENTIONS:
Drug: Cadonilimab — a PD-1/CTLA-4 dual antibody
Radiation: Low-dose radiotherapy — Low-dose radiation
Radiation: SBRT — selected leisions to treat with stereotactic radiotherapy
  Arms: Hybrid RT
Drug: Capecitabine — Capecitabine metronomic chemotherapy
  Arms: Metronomic chemotherapy and LDRT

SUMMARY:
Currently, there is a lack of high-quality clinical evidence for subsequent treatment options for recurrent/metastatic head and neck squamous cell carcinoma (HNSCC) after first-line treatment, especially for subsequent treatment after first-line therapy combined with PD-1 inhibitors. Increasing evidence suggests that low-dose radiation (LDRT) can reshape the tumor microenvironment.Cadonilimab is a bispecific antibody that specifically binds to CTLA-4 and PD-1 proteins in the human body.

Considering that low-dose radiotherapy and cadonilimab both have immunomodulatory effects, this study intends to select recurrent metastatic HNSCC patients who have failed first-line and above treatment to explore the safety and efficacy of cadonilimab combined with low-dose radiotherapy.

DETAILED DESCRIPTION:
Currently, there is a lack of high-quality clinical evidence for subsequent treatment options for recurrent/metastatic head and neck squamous cell carcinoma (HNSCC) after first-line treatment, especially for subsequent treatment after first-line therapy combined with PD-1 inhibitors. Increasing evidence suggests that low-dose radiation (LDRT) can reshape the tumor microenvironment, polarize macrophages towards M1, and M1 macrophages secrete chemokines to promote the recruitment of effector T cells while inducing vascular normalization.

Cadonilimab is a bispecific antibody that specifically binds to CTLA-4 and PD-1 proteins in the human body. It is the first approved PD-1/CTLA-4 bispecific antibody. In June 2022, cadonilimab was approved by the NMPA for the treatment of recurrent or metastatic cervical cancer patients after platinum-based chemotherapy failure. The drug is currently undergoing clinical trials for other types of cancers, including non-small cell lung cancer, hepatocellular carcinoma, gastric cancer, esophageal cancer, and nasopharyngeal cancer.

In view of the subsequent treatment strategies for recurrent metastatic HNSCC after first-line treatment progress, there is still a lack of high-level evidence-based medical evidence to confirm the best recommendation for subsequent treatment. Considering that low-dose radiotherapy and cadonilimab both have immunomodulatory effects, this study intends to select recurrent metastatic HNSCC patients who have failed first-line and above treatment to explore the safety and efficacy of cadonilimab combined with low-dose radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who signed the informed consent and were willing to complete the study according to the protocol;
2. Aged ≥18 years and ≤75 years;
3. Histologically confirmed head and neck squamous cell carcinoma or nasopharyngeal carcinoma;
4. Patients with recurrent and metastatic head and neck squamous cell carcinoma or nasopharyngeal carcinoma, with progression on first-line treatment or above; or locally advanced head and neck squamous cell carcinoma or nasopharyngeal carcinoma, with recurrence and metastasis within 6 months after radical radiotherapy;
5. For patients with locally recurrent head and neck squamous cell carcinoma or nasopharyngeal carcinoma, those who are not suitable for local treatment after multidisciplinary evaluation of head and neck tumors;
6. At least one measurable lesion before treatment, that is, meeting the "measurable lesion" requirement in the RECIST 1.1 standard;
7. Expected survival period>3 months;
8. ECOG score 0-2 points;
9. Good organ function: meet the following requirements:

   1. Absolute neutrophil count (ANC) ≥1.5×109/L;
   2. Platelet count ≥100×109/L;
   3. Hemoglobin ≥9g/dL;
   4. Serum albumin ≥2.8g/dL;
   5. Total bilirubin ≤1.5×ULN, ALT, AST and/or ALP ≤3×ULN;
   6. Serum creatinine ≤1.5×ULN and creatinine clearance ≥60 mL/min (Cockcroft-Gault, see Appendix 3);
   7. Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤1.5× ULN (screening is allowed for patients who are taking stable doses of anticoagulant therapy such as low molecular weight heparin or warfarin and whose INR is within the expected therapeutic range of the anticoagulant);
10. Patients with hepatitis B virus (HBV) infection and inactive/asymptomatic HBV carriers, or patients with chronic or active HBV, will be allowed to enroll if HBV DNA <500 IU/mL (or 2500 copies/mL) at screening. Patients with positive hepatitis C antibodies will be allowed to enroll if HCV-RNA is negative at screening.
11. Women of childbearing age need to have a negative urine or serum pregnancy test result within ≤7 days before treatment. And use a medically approved contraceptive method (such as intrauterine device, birth control pills or condoms) during the study treatment, at least 3 months after the last use of cadonilimab, and at least 6 months after the last use of chemotherapy;
12. Male subjects who are not sterilized must be willing to use a medically approved contraceptive method (such as intrauterine device, birth control pills or condoms) during the study treatment, at least 3 months after the last use of cadonilimab, and at least 6 months after the last use of chemotherapy.

Exclusion Criteria:

1. Patients who have received anti-CTLA-4 antibodies, or any other antibodies or drugs targeting T cell co-stimulation or checkpoint pathways, or small molecule tyrosine kinase inhibitors, including lenvatinib, anlotinib, apatinib, etc.;
2. Patients with symptoms of spinal cord compression, risk of pathological fracture, or emergency surgery and/or radiotherapy due to other medical needs;
3. Patients with a history of gastrointestinal perforation and/or fistula within 6 months before enrollment (if the gastrointestinal perforation or fistula has been surgically removed, enrollment is allowed);
4. Patients with necrotic lesions within 4 weeks before enrollment, or tumors directly invading the trachea, bronchus, esophagus, or arteries, and who are judged by the investigator to have a risk of major bleeding;
5. Patients with other malignant tumors in the past or at the same time (except for malignant tumors that have been cured and have survived without cancer for more than 3 years, such as basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary thyroid carcinoma);
6. Uncontrolled clinical symptoms or diseases of the heart, such as: a. NYHA heart failure of grade II or above; b. Unstable angina pectoris; c. Myocardial infarction within 1 year; d. Patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
7. Received any of the following treatments:

   1. Received any research drug within 4 weeks before the first use of the study drug;
   2. Enrolled in another clinical study at the same time, unless it is an observational (non-interventional) clinical study;
   3. Subjects who need to be given corticosteroids (daily prednisone equivalent dose of >10 mg) or other immunosuppressants for systemic treatment within 2 weeks before the first use of the study drug, except for the use of corticosteroids for local inflammation and prevention of allergies, nausea and vomiting. Other special cases need to be communicated with the investigator. In the absence of active autoimmune diseases, inhaled or topical steroids and adrenocortical hormone replacement at a dose of >10 mg/day prednisone are allowed;
   4. Patients who have received anti-tumor vaccines or have received vaccines (including live vaccines or inactivated vaccines) within 4 weeks before the first administration of the study drug;
   5. Patients who have undergone major surgery or severe trauma within 4 weeks before the first use of the study drug;
8. The toxicity of previous anti-tumor treatment has not recovered to ≤CTCAE grade 1 (except for sequelae of alopecia and neurotoxicity related to previous platinum treatment) or the level specified by the inclusion/exclusion criteria;
9. Severe infection (CTCAE>2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, bacteremia, infectious complications, etc. requiring hospitalization; baseline chest imaging examinations indicate active lung inflammation, symptoms and signs of infection within 4 weeks of the first use of the study drug, or the need for oral or intravenous antibiotic treatment;
10. Active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); but not including autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone; type 1 diabetes using stable doses of insulin; patients with vitiligo or healed childhood asthma/allergies who do not require any intervention as adults;
11. Patients with a history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation;
12. Patients with a history of interstitial lung disease (excluding radiation pneumonia without steroid treatment) or non-infectious pneumonia;
13. Patients with active pulmonary tuberculosis infection found through medical history or CT examination, or patients with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than 1 year ago but without formal treatment;
14. Subjects with active hepatitis B (HBV DNA ≥500 IU/mL or 2500 copies/mL), hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method);
15. known history of psychotropic drug abuse, alcoholism or drug abuse;
16. pregnant or lactating women;
17. the researcher judges that the subject has other factors that may force him to terminate the study midway, such as other serious diseases (including mental illness) requiring combined treatment, serious abnormal laboratory test values, family or social factors that may affect the safety of the subject or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to two years
  Objective Response Rate (ORR), as assessed by investigators according to RECIST 1.1 criteria. For patients who have received radiotherapy for all lesions, the ORR assessment should be based on the lesions that received SBRT and low-dose radiotherapy. For patients with lesions that did not receive radiotherapy, the ORR assessment should be based on the lesions that received SBRT, low-dose radiotherapy, and those that did not receive radiotherapy

SECONDARY OUTCOMES:
Adverse effect | Up to two years
  Adverse effects (AE) as evaluated by CTCAE 5.0
Disease Control Rate | Up to two years
  Disease Control Rate (DCR), as assessed by investigators according to RECIST 1.1 criteria
Duration of Response | Up to two years
  Duration of Response (DoR), as assessed by investigators according to RECIST 1.1 criteria
Progression-free survival | Up to two years
  Progression-free survival (PFS): from the start of enrollment to the first recorded date of objective tumor progression or death from any cause, whichever occurs first.
Overall survival | Up to two years
  Overall survival (OS): the time from enrollment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Wang, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD unless special request to principal invesitgators with formal applications.

REFERENCES:
- [Background] Keam SJ. Cadonilimab: First Approval. Drugs. 2022 Aug;82(12):1333-1339. doi: 10.1007/s40265-022-01761-9. PMID 35986837
- [Background] Gao X, Xu N, Li Z, Shen L, Ji K, Zheng Z, Liu D, Lou H, Bai L, Liu T, Li Y, Li Y, Fan Q, Feng M, Zhong H, Huang Y, Lou G, Wang J, Lin X, Chen Y, An R, Li C, Zhou Q, Huang X, Guo Z, Wang S, Li G, Fei J, Zhu L, Zhu H, Li X, Li F, Liao S, Min Q, Tang L, Shan F, Gong J, Gao Y, Zhou J, Lu Z, Li X, Li J, Ren H, Liu X, Yang H, Li W, Song W, Wang ZM, Li B, Xia M, Wu X, Ji J. Safety and antitumour activity of cadonilimab, an anti-PD-1/CTLA-4 bispecific antibody, for patients with advanced solid tumours (COMPASSION-03): a multicentre, open-label, phase 1b/2 trial. Lancet Oncol. 2023 Oct;24(10):1134-1146. doi: 10.1016/S1470-2045(23)00411-4. PMID 37797632
- [Background] Herrera FG, Ronet C, Ochoa de Olza M, Barras D, Crespo I, Andreatta M, Corria-Osorio J, Spill A, Benedetti F, Genolet R, Orcurto A, Imbimbo M, Ghisoni E, Navarro Rodrigo B, Berthold DR, Sarivalasis A, Zaman K, Duran R, Dromain C, Prior J, Schaefer N, Bourhis J, Dimopoulou G, Tsourti Z, Messemaker M, Smith T, Warren SE, Foukas P, Rusakiewicz S, Pittet MJ, Zimmermann S, Sempoux C, Dafni U, Harari A, Kandalaft LE, Carmona SJ, Dangaj Laniti D, Irving M, Coukos G. Low-Dose Radiotherapy Reverses Tumor Immune Desertification and Resistance to Immunotherapy. Cancer Discov. 2022 Jan;12(1):108-133. doi: 10.1158/2159-8290.CD-21-0003. Epub 2021 Sep 3. PMID 34479871